CLINICAL TRIAL: NCT03324815
Title: Analgesic Effect Evaluation of Methadone Associated With Morphine for Cancer Pain: Prospective Randomized Study
Brief Title: Methadone Associated With Morphine for Cancer Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Feliciano Contardo Nepomuceno Duarte, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30850414.0.0000.5505
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Cancer
Keywords: Morphine; Methadone; Pain
MeSH Terms: conditions — Neoplasms; Pain | interventions — Morphine; Methadone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morphine- Methadone (Active Comparator): Morphine 5mg/6h plus metadone: 2,5mg/12h
  Interventions: Drug: Morphine; Drug: Methadone
- Morphine (Active Comparator): Morphine: 5mg/6h
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — Pain Treatment
  Other Names: Dimorf
Drug: Methadone — Pain Treatment
  Other Names: Mytedom
  Arms: Morphine- Methadone

SUMMARY:
The study was prospective, randomized. Patients with cancer pain were evaluated, one group receiving methadone with morphine and another group receiving morphine as the only opioid. Pain intensity, total morphine dose and adverse effects were evaluated.

DETAILED DESCRIPTION:
Opioids are the most important analgesics for the relief of cancer pain. In addition tolerance and hyperalgesia may ocurr as a consequence of treatment with these drugs. Medications for pain relief may also cause increased pain. NMDA receptor blockers may prevent or reduce the development of hyperalgesia. Methadone is a weak NMDA receptor antagonist and therefore its association could prevent hyperalgesia. The primary endpoint of the study was whether the administration of low dose methadone associated with morphine promotes better analgesic effect in patients with cancer pain, And secondarily to assess whether there is a reduction in the total dose of opioid needed for pain relief, and whether reduction of the opioid-related adverse effects occurs.

ELIGIBILITY:
Inclusion Criteria:

* Approved by the Ethics Committee
* signed the informed consent
* cancer pain
* starting the WHO thirth analgesic ladder,

Exclusion Criteria:

* cognitive impairment
* psychiatric disease
* illicit drug user
* hypersensitivity to the study drugs
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-08-30 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 3 months
  Total dose of morphine used by the patient

SECONDARY OUTCOMES:
Pain intensity | 3 months
  Measure of pain intensity by verbal numerical rating score (VNRS - zero to 10) where 0 is no pain and 10 is the worst pain imaginable. Values between 0 and 3 mean a good result, between 4 and 6 a poor result and between 7 and 10 a very poor result.

CONTACTS AND LOCATIONS:
Overall Officials: Rioko K Sakata, MD; PhD, Principal Investigator — Universidade Federal de São Paulo
Locations (1):
- Rioko K Sakata, São Paulo, Brazil

REFERENCES:
- [Derived] Duarte FCN, Ferraro LHDC, Ferreira A, Sakata RK. A Randomized Controlled Trial Evaluating the Analgesic Effect of the Combination of Methadone With Morphine for Cancer Related Pain. Clin J Pain. 2021 Sep 1;37(9):664-668. doi: 10.1097/AJP.0000000000000959. PMID 34265791